CLINICAL TRIAL: NCT06887855
Title: Enhancing Post-Stroke Dysphagia Rehabilitation Via the Synergistic Effects of Neuromuscular Electrical Stimulation, Neuromuscular Taping, and Swallowing Exercises: a Randomized Controlled Trial
Brief Title: Enhancing Post-Stroke Dysphagia Rehabilitation
Acronym: Not exist
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Ibrahim Mohammed Abdul Fattah Al Ayaseh, Speech-Language Pathology Supervisor, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-23-242; Not exist (Other Grant/Funding Number: Hamad Medical Corporation)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Dysphagia After Stroke
Keywords: post-stroke; dysphagia; combined rehabilitation; neuromuscular electrical stimulation; kinesiology taping; neuromuscular taping; chin tuck against resistance; expiratory muscle strength training
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: The study includes 3 intervention groups.
Masking Description: The outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Participants will receive neuromuscular electrical stimulation + swallowing exercises ( chin tuck against resistance + expiratory muscle strength training)
  Interventions: Procedure: Neuromuscular Electrical Stimulation; Procedure: Swallowing exercise (Expiratory Muscle Strength Training); Procedure: Swallowing exercise (Chin Tuck Against Resistance)
- Group B (Experimental): Participants will receive neuromuscular taping + swallowing exercises (chin tuck against resistance + expiratory muscle strength training)
  Interventions: Procedure: Neuromuscular Taping; Procedure: Swallowing exercise (Expiratory Muscle Strength Training); Procedure: Swallowing exercise (Chin Tuck Against Resistance)
- Group C (Experimental): Participants will receive neuromuscular electrical stimulation + neuromuscular taping + swallowing exercises (chin tuck against resistance + expiratory muscle strength training)
  Interventions: Procedure: Neuromuscular Electrical Stimulation; Procedure: Neuromuscular Taping; Procedure: Swallowing exercise (Expiratory Muscle Strength Training); Procedure: Swallowing exercise (Chin Tuck Against Resistance)

INTERVENTIONS:
Procedure: Neuromuscular Electrical Stimulation — NMES is a modality for stimulating muscles through electrical pulses, is used widely in the rehabilitation of stroke patients with pharyngeal dysphagia. It reinforces the strength of the muscles for swallowing and smooths the swallowing reflex through sensory stimulation. Clinically, NMES is applied to depolarize nerve fibers at the point of engagement, involving muscle contraction (Park et al. 2019). NMES includes the placement of electrical stimuli to the skin around the face and neck through surface electrodes. Stimulation intensity can be diverse depending on the treatment objectives. Low-intensity (sensory) NMES lets patients feel the tingling sensation on the skin, whereas high-intensity (motor) NMES can stimulate muscle contractions (Cheng et al. 2022).
  Arms: Group A; Group C
Procedure: Neuromuscular Taping — NMT is similar to kinesiology taping but specifically focuses on neuromuscular re-education and it is a commonly used therapy approach for various neuromuscular problems. The neuromuscular tape can be easily applied to skeletal muscles to induce or inhibit muscle activity and to support the stabilization of structures such as joints and ligaments. The elasticity and adhesion properties of NMT can be used to restrain the anterior-upward movement of the hyolaryngeal complex during spontaneous swallowing. This effect increases the load on the suprahyoid muscles and consequently, the patient spends more effort to overcome this movement while swallowing. Resistance exercises provided with NMT activate the suprahyoid muscle and contractions for the muscles of the tongue.
  Arms: Group B; Group C
Procedure: Swallowing exercise (Expiratory Muscle Strength Training) — IN EMST the patients blow into a one-way spring-loaded apparatus calibrated to a percentage of maximum expiratory pressure until the valve opens with adequate effort. Four to eight weeks of EMST exercises increased the maximum expiratory pressure (MEP), maximum hyoid displacement, suprahyoid muscle action, and swallowing safety in patients with amyotrophic lateral sclerosis, stroke, and neck cancer.
Procedure: Swallowing exercise (Chin Tuck Against Resistance) — CTAR exercise is performed by an inflatable 12 cm rubber ball. The patients are directed to sit upright on a chair and hold the rubber ball between the base of the chin and the manubrium sterna. This exercise is composed of isometric and isotonic movements. The isometric movement will be performed for 10 seconds, whereas the isokinetic movement will be successively repeated 10 times to strengthen the suprahyoid and infrahyoid muscles (Kagaya & Inamoto, 2022).

SUMMARY:
The goal of this clinical trial is to investigate the effects of a combined swallowing intervention (Neuromuscular Electrical Stimulation (NMES) + Neuromuscular Taping (NMT) + swallowing exercises) on swallowing function and quality of life in post-stroke dysphagia patients. The main questions it aims to answer are:

• Does the combination of swallowing exercises, NMES & NMT have a greater improvement in dysphagia rehabilitation when compared to either NMES or NMT alone? Researchers will compare the effects of intervention between the three groups (NMES and swallowing exercises, NMT and swallowing exercises, and NMES with NMT and swallowing exercises).

Participants will:

* Receive a combined dysphagia rehabilitation comprised of swallowing exercises, Neuromuscular Electrical stimulation, and/or Neuromuscular Taping.
* Visit the clinic once every 5 days a week for 10 therapy sessions.
* Undergo baseline and post-intervention evaluation procedures.

DETAILED DESCRIPTION:
This proposed study will be conducted using a prospective, three-group, randomized controlled trial. The participants for this study will be recruited from the post-acute and rehabilitation units who are diagnosed with post-stroke dysphagia at Hamad Medical Corporation hospitals in the State of Qatar.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 75 years old,
* Diagnosed with swallowing disorders between one day and six months post-stroke,
* Able to attend 10 therapy sessions,
* Have never received any swallowing treatment before participating in this study.

Exclusion Criteria:

* Post-stroke patients with severe cognitive impairment,
* Patients who have swallowing disorders due to other etiologies,
* Patients who need traditional swallowing therapy other than Expiratory Muscle Strength Training (EMST) and Chin Tuck Against Resistance (CTAR). - Skin disorders in the submental area and anterior neck,
* Medical conditions that may affect participation,
* A defibrillator and use precision electrical biomedical devices (e.g. pacemaker, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male/female
Enrollment: 10 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale (PAS) score | Pre-intervention: "Baseline" or "Day 1". Post-intervention: immediately after the intervention, up to 15 days of start the intervention.
  It is an 8-point ordinal scale, with 1 representing the least and 8 representing the highest or most severe score. PAS scores are multidimensional, i.e., include several observations within each score: (1) depth of airway invasion (material above, contacting, or below the level of vocal folds; (2) whether or not there is material remaining after the swallow (ejected, not ejected); and (3) the patient's response to material present in the airway (effort to clear the material)
Dysphagia Handicap Index | Pre-intervention: "Baseline" or "Day 1". Post-intervention: immediately after the intervention, up to 15 days of start the intervention.
  Dysphagia Handicap Index is comprised of a 25-item self-administered questionnaire. It is an instrument for measuring the handicapping impact of swallowing disorder on the physical, functional, and emotional facets of individuals' lives.
  Respondents replied never, sometimes, or always to each statement and rated their self-perceived dysphagia severity on a 7-point equal-appearing interval scale. 1 indicates normal swallowing and 7 indicates server swallowing problem.
surface Electromyography (sEMG) | Pre-intervention: "Baseline" or "Day 1". Post-intervention: immediately after the intervention, up to 15 days of start the intervention.
  Surface EMG biofeedback is typically implemented by placing surface electrodes over a patient's under-chin area or submental muscles to observe the changes in muscle actions during swallowing. The recorded signals are processed and converted into a visual demonstration or auditory prompt. The participants' swallowing muscles (suprahyoid) performance will be measured using the maximum work parameter to compare each participant's performance per- and post- intervention.

SECONDARY OUTCOMES:
DYSPHAGIA OUTCOME SEVERITY SCALE (DOSS) | Pre-intervention: "Baseline" or "Day 1". Post-intervention: immediately after the intervention, up to 15 days of start the intervention.
  DOSS is a simple, easy-to-use, 7-point scale developed to systematically rate the functional severity of dysphagia based on objective assessment and make recommendations for diet level, independence level, and type of nutrition.
Hyoid bone displacement | Pre-intervention: "Baseline" or "Day 1". Post-intervention: immediately after the intervention, up to 15 days of start the intervention.
  The physiology of swallowing involves many biomechanical processes, such as displacement of the hyoid bone, which is an important part of protecting the airway and the opening of the upper esophageal sphincter. The displacement of the hyoid bone will be measured based on the videofluoroscopic swallow study.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Mohammad Alayaseh, M.Sc. _ SLP, Study Chair — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Baladīyat ad Dawḩah, Qatar

IPD SHARING:
Plan to Share IPD: No
Data sharing requires permission from the Qatar Ministry of Public Health. Any request for data requisition can be made to the Medical Research Center (MRC) at Hamad Medical Corporation Qatar, which will seek legal permission from the Ministry of Public Health before sharing the data.

REFERENCES:
- [Background] Xia W, Zheng C, Lei Q, Tang Z, Hua Q, Zhang Y, Zhu S. Treatment of post-stroke dysphagia by vitalstim therapy coupled with conventional swallowing training. J Huazhong Univ Sci Technolog Med Sci. 2011 Feb;31(1):73-76. doi: 10.1007/s11596-011-0153-5. Epub 2011 Feb 19. PMID 21336727
- [Background] Wang Y, Li X, Sun C, Xu R. Effectiveness of kinesiology taping on the functions of upper limbs in patients with stroke: a meta-analysis of randomized trial. Neurol Sci. 2022 Jul;43(7):4145-4156. doi: 10.1007/s10072-022-06010-1. Epub 2022 Mar 26. PMID 35347525
- [Background] Teo, J. T., Chin, Y. L., & Wong, M. L. (2021). Dysphagia management in post-stroke patients: The role of combined interventions. Stroke Research and Treatment, 2021, 4520345. https://doi.org/10.1155/2021/4520345
- [Background] Tarihci Cakmak E, Sen EI, Doruk C, Sen C, Sezikli S, Yaliman A. The Effects of Neuromuscular Electrical Stimulation on Swallowing Functions in Post-stroke Dysphagia: A Randomized Controlled Trial. Dysphagia. 2023 Jun;38(3):874-885. doi: 10.1007/s00455-022-10512-7. Epub 2022 Aug 20. PMID 35986170
- [Background] Tan Z, Wei X, Tan C, Wang H, Tian S. Effect of neuromuscular electrical stimulation combined with swallowing rehabilitation training on the treatment efficacy and life quality of stroke patients with dysphagia. Am J Transl Res. 2022 Feb 15;14(2):1258-1267. eCollection 2022. PMID 35273727
- [Background] Sproson L, Pownall S, Enderby P, Freeman J. Combined electrical stimulation and exercise for swallow rehabilitation post-stroke: a pilot randomized control trial. Int J Lang Commun Disord. 2018 Mar;53(2):405-417. doi: 10.1111/1460-6984.12359. Epub 2017 Dec 30. PMID 29288590
- [Background] Silva APD, Carvalho ARR, Sassi FC, Andrada E Silva MA. The taping method effects on the trapezius muscle in healthy adults. Codas. 2019 Oct 17;31(5):e20180077. doi: 10.1590/2317-1782/20192018077. eCollection 2019. English, Portuguese. PMID 31644716
- [Background] Silbergleit AK, Schultz L, Jacobson BH, Beardsley T, Johnson AF. The Dysphagia handicap index: development and validation. Dysphagia. 2012 Mar;27(1):46-52. doi: 10.1007/s00455-011-9336-2. Epub 2011 Mar 20. PMID 21424584
- [Background] Propp R, Gill PJ, Marcus S, Ren L, Cohen E, Friedman J, Mahant S. Neuromuscular electrical stimulation for children with dysphagia: a systematic review. BMJ Open. 2022 Mar 25;12(3):e055124. doi: 10.1136/bmjopen-2021-055124. PMID 35338059
- [Background] Park JW, Kim Y, Oh JC, Lee HJ. Effortful swallowing training combined with electrical stimulation in post-stroke dysphagia: a randomized controlled study. Dysphagia. 2012 Dec;27(4):521-7. doi: 10.1007/s00455-012-9403-3. Epub 2012 Mar 24. PMID 22447240
- [Background] Park JS, Hwang NK, Kim HH, Lee G, Jung YJ. Effect of neuromuscular electrical stimulation combined with effortful swallowing using electromyographic biofeedback on oropharyngeal swallowing function in stroke patients with dysphagia: A pilot study. Medicine (Baltimore). 2019 Nov;98(44):e17702. doi: 10.1097/MD.0000000000017702. PMID 31689798
- [Background] Meng P, Zhang S, Wang Q, Wang P, Han C, Gao J, Yue S. The effect of surface neuromuscular electrical stimulation on patients with post-stroke dysphagia. J Back Musculoskelet Rehabil. 2018;31(2):363-370. doi: 10.3233/BMR-170788. PMID 29278871
- [Background] Matos KC, de Oliveira VF, de Oliveira PLC, Carvalho FA, de Mesquita MRM, da Silva Queiroz CG, Marques LM, Lima DLN, Carvalho FMM, Braga-Neto P. Combined conventional speech therapy and functional electrical stimulation in acute stroke patients with dyphagia: a randomized controlled trial. BMC Neurol. 2022 Jun 22;22(1):231. doi: 10.1186/s12883-022-02753-8. PMID 35733098
- [Background] Marcus S, Friedman JN, Lacombe-Duncan A, Mahant S. Neuromuscular electrical stimulation for treatment of dysphagia in infants and young children with neurological impairment: a prospective pilot study. BMJ Paediatr Open. 2019 Jan 23;3(1):e000382. doi: 10.1136/bmjpo-2018-000382. eCollection 2019. PMID 30740545
- [Background] Lin CL, Wu WT, Chang KV, Lin HY, Chou LW. Application of Kinesio Taping method for newborn swallowing difficultly: A case report and literature review. Medicine (Baltimore). 2016 Aug;95(31):e4458. doi: 10.1097/MD.0000000000004458. PMID 27495080
- [Background] Li L, Li Y, Huang R, Yin J, Shen Y, Shi J. The value of adding transcutaneous neuromuscular electrical stimulation (VitalStim) to traditional therapy for post-stroke dysphagia: a randomized controlled trial. Eur J Phys Rehabil Med. 2015 Feb;51(1):71-8. Epub 2014 Jul 23. PMID 25052012
- [Background] Jung YJ, Kim HJ, Choi JB, Park JS, Hwang NK. Effect of Dysphagia Rehabilitation Using Kinesiology Taping on Oropharyngeal Muscle Hypertrophy in Post-Stroke Patients: A Double Blind Randomized Placebo-Controlled Trial. Healthcare (Basel). 2020 Oct 19;8(4):411. doi: 10.3390/healthcare8040411. PMID 33086705
- [Background] Jing, Q., Yang, X., & Reng, Q. (2016). Effect of neuromuscular electrical stimulation in patients with post-stroke dysphagia. Medical Science and Technology, 57, 1-5. https://doi.org/10.12659/MST.895042
- [Background] Howard MM, Block ES, Mishreki D, Kim T, Rosario ER. The Effect of Sensory Level Versus Motor Level Electrical Stimulation of Pharyngeal Muscles in Acute Stroke Patients with Dysphagia: A Randomized Trial. Dysphagia. 2023 Jun;38(3):943-953. doi: 10.1007/s00455-022-10520-7. Epub 2022 Sep 20. PMID 36127447
- [Background] Gulec A, Albayrak I, Erdur O, Ozturk K, Levendoglu F. Effect of swallowing rehabilitation using traditional therapy, kinesiology taping and neuromuscular electrical stimulation on dysphagia in post-stroke patients: A randomized clinical trial. Clin Neurol Neurosurg. 2021 Dec;211:107020. doi: 10.1016/j.clineuro.2021.107020. Epub 2021 Nov 6. PMID 34781221
- [Background] Du B, Li Y, Zhang B, Zhao W, Zhou L. Effect of neuromuscular electrical stimulation associated with swallowing-related muscle training for post-stroke dysphagia: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2021 Mar 19;100(11):e25108. doi: 10.1097/MD.0000000000025108. PMID 33725989
- [Background] Coman LM, Cardell EA, Richards JA, Mahon A, Lawrie MD, Ware RS, Weir KA. Videofluoroscopic swallow study training for radiologists-in-training: a survey of practice and training needs. BMC Med Educ. 2022 Nov 7;22(1):762. doi: 10.1186/s12909-022-03799-5. PMID 36344980
- [Background] Chen, P., Zhang, X., Li, Y., & Wang, T. (2020). The impact of dysphagia on quality of life in post-stroke patients: A systematic review and meta-analysis. Journal of Stroke and Cerebrovascular Diseases, 29(2), 145-153. https://doi.org/10.1016/j.jstrokecerebrovasdis.2019.12.011
- [Background] Cheng I, Hamad A, Sasegbon A, Hamdy S. Advances in the Treatment of Dysphagia in Neurological Disorders: A Review of Current Evidence and Future Considerations. Neuropsychiatr Dis Treat. 2022 Oct 14;18:2251-2263. doi: 10.2147/NDT.S371624. eCollection 2022. PMID 36268265
- [Background] Carnaby GD, LaGorio L, Silliman S, Crary M. Exercise-based swallowing intervention (McNeill Dysphagia Therapy) with adjunctive NMES to treat dysphagia post-stroke: A double-blind placebo-controlled trial. J Oral Rehabil. 2020 Apr;47(4):501-510. doi: 10.1111/joor.12928. Epub 2020 Jan 19. PMID 31880338
- [Background] Byeon H. Combined Effects of NMES and Mendelsohn Maneuver on the Swallowing Function and Swallowing-Quality of Life of Patients with Stroke-Induced Sub-Acute Swallowing Disorders. Biomedicines. 2020 Jan 12;8(1):12. doi: 10.3390/biomedicines8010012. PMID 31940930
- [Background] Banda KJ, Chu H, Kang XL, Liu D, Pien LC, Jen HJ, Hsiao SS, Chou KR. Prevalence of dysphagia and risk of pneumonia and mortality in acute stroke patients: a meta-analysis. BMC Geriatr. 2022 May 13;22(1):420. doi: 10.1186/s12877-022-02960-5. PMID 35562660